CLINICAL TRIAL: NCT06941558
Title: INFINITY™ With ADAPTIS™ and EVERLAST™ Technology Total Ankle Replacement Follow-up
Brief Title: The UK ADAPTIS Study
Acronym: UK ADAPTIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHCT0494
Record Dates: First submitted 2025-03-27; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Total Ankle Replacement; Total Ankle Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- INFINITY™ with ADAPTIS™ and EVERLAST™ (Other): INFINITY™ with ADAPTIS™ and EVERLAST™ technology with Poly Insert for patients requiring primary TAA/TAR.
  Interventions: Device: INFINITY™ with ADAPTIS™ and EVERLAST™

INTERVENTIONS:
Device: INFINITY™ with ADAPTIS™ and EVERLAST™ — The INFINITY™ with ADAPTIS™ and EVERLAST™ ankle replacement system is a development of the Infinity ankle implant, designed to attach to the bone better and to wear out more slowly.

SUMMARY:
An ankle replacement procedure consists of replacing the worn-out joint surfaces of the ankle with metal and plastic components that are shaped to allow continued movement of the ankle. There are several different types of ankle replacement available. Infinity ankle implants are already routinely used in NHS hospitals. The INFINITY™ with ADAPTIS™ and EVERLAST™ ankle replacement system is a development of the Infinity ankle implant, designed to attach to the bone better and to wear out more slowly.

The purpose of the UK ADAPTIS™ Study is to assess the performance and function of the newly introduced INFINITY™ with ADAPTIS™ and EVERLAST™ technology Total Ankle System for total ankle replacement (TAR) or arthroplasty (TAA) and EVERLAST™ Poly Insert that modernises and streamlines Stryker's TAA/TAR portfolio.

UK ADAPTIS is a prospective multi-centre cohort series of INFINITY™ with ADAPTIS™ and EVERLAST™ Technology with Poly Insert for patients requiring primary total ankle replacement (TAR) i.e. Total Ankle Arthroplasty (TAA).

Patients meeting the criteria for the study will be asked to enrol by providing written informed consent.

The patients will be monitored clinically by post-operative follow-up examinations and Patient reported outcome measures (PROMs) (Manchester Oxford Foot & Ankle Questionnaire (MOXFQ), Ankle Osteoarthritis Scale (AOS), EQ5D-5L).

Intended use:

It is intended to give a patient limited mobility by reducing pain, restoring alignment, and replacing flexion and extension movement in the ankle joint.

Indications for use:

* Patients with ankle joints damaged by severe rheumatoid, post-traumatic, or degenerative arthritis.
* Patients with a failed previous ankle surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female over the age of 21 years with a diagnosis of end stage ankle arthritis and requiring primary TAA/TAR and is suitable for the use of the ADAPTIS TAA/TAR
2. Patients who are physically and mentally willing and able to comply with the post-operative follow-ups and an appropriate rehabilitation schedule.
3. Patient can understand and provide written consent.

Exclusion Criteria:

1. Patients with previous ankle arthrodesis or Patients who require revision of previously implanted TAA/TAR.
2. Any patients presenting with clinically relevant conditions prior to implantation, that would contraindicate implantation of a TAA/TAR

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Functional Status | 2 years
  Functional status using MOXFQ (Manchester-Oxford Foot Questionnaire). The MOXFQ is scored on a 0-100 scale, where higher scores indicate more severe problems.
Device Survivorship | 2 years
  Device survivorship, assessed by tracking revision rates
Device Survivorship | 2 years
  Device survivorship, assessed by tracking re-operations
Device Survivorship | 2 years
  Device survivorship, assessed by adverse events

SECONDARY OUTCOMES:
Pain and Disability | Up to 5 years post-op
  Pain and disability assessed using AOS (Ankle Osteoarthritis Scale) questionnaire. A higher score on the AOS reflects greater pain, functional limitations, and a generally poorer overall ankle-related health status.
Pain and Disability | Up to 5 years post-op
  Pain and disability assessed using MOXFQ (Manchester-Oxford Foot Questionnaire). The MOXFQ is scored on a 0-100 scale, where higher scores indicate more severe problems.
Pain and Disability | Up to 5 years post-op
  Pain and disability assessed using a specific health-related quality of life questionnaire (EQ5D-5L)

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria Healthcare NHS Foundation Trust, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that a publication of the anonymous study results will be compiled and submitted to a peer-reviewed journal. The CI of the study will have the responsibility of being primary author of such publications.
  The study will be registered in the ISRCTN Trial Register and/or in clinicaltrials.gov by the CI.